CLINICAL TRIAL: NCT04454788
Title: Extending the Time Window for Tenecteplase by Effective Reperfusion of PeNumbrAL Tissue in Patients with Large Vessel Occlusion
Brief Title: Extending the Time Window for Tenecteplase by Effective Reperfusion in Patients with Large Vessel Occlusion
Acronym: ETERNAL-LVO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Loss of equipoise in the 0-4.5h population which comprised the majority of ETERNAL-LVO trial recruitment due to publication of other trials demonstrating efficacy of tenecteplase vs alteplase in the 0-4.5h time window.
Sponsor: University of Melbourne (Other)
Collaborators: Professor Mark Parsons (Unknown)
Responsible Party: Principal Investigator, Bruce Campbell, Prof, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.125
Record Dates: First submitted 2020-06-16; First posted 2020-07-02 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous tenecteplase (TNK) (Experimental): Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds).
  Interventions: Drug: Tenecteplase
- Intravenous tissue plasminogen activator (tPA) (Active Comparator): Patients will receive standard of care (no intravenous thrombolytic treatment or intravenous alteplase 0.9mg/kg at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour.
  Interventions: Drug: Standard Care (which may include intravenous Alteplase)

INTERVENTIONS:
Drug: Tenecteplase — Genetically modified tissue plasminogen activator at a dose of 0.25mg/kg given as intravenous bolus over 5-10 seconds
  Arms: Intravenous tenecteplase (TNK)
Drug: Standard Care (which may include intravenous Alteplase) — Patients will receive standard care which may include intravenous alteplase at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour.
  Arms: Intravenous tissue plasminogen activator (tPA)

SUMMARY:
Patients presenting to the emergency department with an acute ischemic stroke due to a large vessel occlusion eligible for thrombectomy and target mismatch on computed tomography perfusion imaging within 24 hours of onset will be assessed determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomised using a central computerised allocation process to either standard of care (no intravenous thrombolytic treatment or intravenous alteplase 0.9mg/kg) or tenecteplase before undergoing intra-arterial clot retrieval. The trial is prospective, randomised, open-label, blinded endpoint (PROBE) design.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute hemispheric ischemic stroke with onset (or the time they last known to be well) within 24 hours.
* Patient's age is ≥18 years.
* Premorbid mRS <3, with a concurrent assessment of whether the patient was able, immediately prior to the stroke, to: 1) Drive, or (if never drives) perform own Domestic duties, and 2) Shop for themselves, and 3) Bank/do their own finances (i.e. Drive/Domestic, Bank, Shop = DBS +ve). Need to be DBS +ve to be study eligible.
* Presence of a vessel occlusion on CTA or MRA. LVO will be defined as 'potentially retrievable' thrombus at one or more of the following sites: intracranial internal carotid (ICA), middle cerebral artery (MCA) first segment (M1), proximal middle cerebral artery second segment (M2) or isolated/tandem occlusion of the extracranial ICA. Patients with an extracranial ICA stenosis and occlusion are also eligible.
* Presence of 'target mismatch' on automated perfusion CT (CTP) or diffusion-perfusion MRI software defined as an ischemic core of <70mL, penumbra of >20mL and an ischemic core to perfusion lesion ratio of >1.8

Exclusion Criteria:

* Intracranial hemorrhage (ICH) or other diagnosis (e.g. tumor).
* Basilar Artery occlusion.
* Extensive early ischemic change (hypodensity on NCCT or high signal on DWI-MRI) or early ischemic change outside the perfusion lesion that invalidates mismatch criteria.
* Pre-stroke mRS score of > 2 (indicating significant previous disability) or DBS -ve.
* Any terminal illness such that patient would not be expected to survive more than 1 year
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
* Pregnant women.
* Other standard contraindications to thrombolysis.
* Minor stroke symptoms, or major stroke symptoms rapidly improving
* Clinical presentation suggesting subarachnoid haemorrhage
* Known bleeding diasthesis and/or platelet count <100,000 or taking warfarin with INR > 1.7.
* Patients who have received heparin within 48 hours must have normal aPTT.
* Major surgery or serious trauma within 14 days, serious head trauma within 3 months.
* GI or urinary tract haemorrhage within last 21 days
* Arterial puncture at a non-compressible site or lumbar puncture within 7 days
* Systolic BP > 185, diastolic BP > 110mmHg
* Clinical stroke within 3 months or history of ICH
* Unable to gain consent from patient or person responsible
* Known severe renal impairment (GFR < 15mls/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 (no disability) or return to baseline mRS | 90 days
  Modified Rankin Scale (mRS) 0-1 (no disability) or return to baseline mRS (if baseline premorbid mRS =2) at 90 days

SECONDARY OUTCOMES:
Early clinical improvement | 24 hours
  Reduction in National Institutes of Health Stroke Scale (NIHSS) score of ≥8 points at 24 hours or reaching NIHSS 0-1
Modified Rankin Scale (mRS) 0-2 (functional independence) | 90 days
  Modified Rankin Scale (mRS) 0-2 (functional independence) at 90 days
Substantial reperfusion at initial angiographic assessment | initial angiography within 24 hours of stroke onset
  Proportion of patients with >50% reperfusion of the affected vascular territory (mTICI 3b/3) on initial digital subtraction angiography prior to thrombectomy
Symptomatic intracerebral hemorrhage (sICH) | 24 hours post-randomization
  sICH defined as parenchymal hematoma type 2 (PH2) - blood clot occupying >30% of the infarcted territory with substantial mass effect
Death due to any cause | 90 days
Modified Rankin Scale (mRS) 5-6 | 90 days
  Poor functional outcome of death or requirement for fulltime nursing care
Successful reperfusion at 24 hours | 24 hours
  Reperfusion (defined as >90% and >50% reduction in perfusion lesion volume)
Infarct growth | 24 hours
  Increase in the volume of irreversibly injured brain between pre-treatment and 24 hour imaging
Recanalization | 24 hours
  Change in vessel patency between pre-treatment and 24h imaging (CT or MR angiography)

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yogendrakumar V, Campbell BCV, Churilov L, Garcia-Esperon C, Choi PMC, Cordato DJ, Dhimal N, Olenko L, Guha P, Sharma G, Chen C, McDonald A, Thijs V, Mamun A, Dos Santos A, Balabanski AH, Kleinig TJ, Butcher KS, Devlin MJ, O'Rourke F, Donnan GA, Davis SM, Levi CR, Ma H, Parsons MW; ETERNAL-LVO Investigators. Efficacy of Tenecteplase in Large Vessel Occlusion Stroke Within 24 Hours of Symptom Onset: The ETERNAL-LVO Randomized Controlled Trial. Stroke. 2025 Dec;56(12):3332-3341. doi: 10.1161/STROKEAHA.125.052511. Epub 2025 Sep 10. PMID 40927857
- [Derived] Yogendrakumar V, Campbell BC, Churilov L, Garcia-Esperon C, Choi PM, Cordato DJ, Guha P, Sharma G, Chen C, McDonald A, Thijs V, Mamun A, Dos Santos A, Balabanski AH, Kleinig TJ, Butcher KS, Devlin MJ, O'Rourke F, Donnan GA, Davis SM, Levi CR, Ma H, Parsons MW. Extending the time window for tenecteplase by effective reperfusion of penumbral tissue in patients with large vessel occlusion: Rationale and design of a multicenter, prospective, randomized, open-label, blinded-endpoint, controlled phase 3 trial. Int J Stroke. 2025 Mar;20(3):367-372. doi: 10.1177/17474930241308660. Epub 2024 Dec 31. PMID 39654273